CLINICAL TRIAL: NCT01237093
Title: Developing Biomarkers of Dietary Intake
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 999911018; 11-DK-N018
Record Dates: First submitted 2010-11-06; First posted 2010-11-09 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-07-25

CONDITIONS: Diet Therapy; Healthy Volunteers
Keywords: Fish Diet; Meat Diet; Biomarkers; Stable Isotopes; Dietary Intake
MeSH Terms: interventions — In Situ Hybridization, Fluorescence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 1. Meat, no fish or soda (Experimental): weight maintaining diet with meat but no fish or soda for 12 weeks
  Interventions: Other: 1. Meat, no fish or soda
- 2. Meat and soda, no fish (Experimental): weight maintaining diet with meat and soda but no fish for 12 weeks
  Interventions: Other: 2. Meat and soda, no fish
- 4. Meat and fish and soda (Experimental): weight maintaining diet with meat, fish, and soda for 12 weeks
  Interventions: Other: 4. Meat and fish and soda
- 5. Fish, no meat or soda (Experimental): weight maintaining diet with meat, fish, and soda for 12 weeks
  Interventions: Other: 5. Fish, no meat or soda
- 6. Fish and soda, no meat (Experimental): weight maintaining diet with fish and soda but no meat for 12 weeks
  Interventions: Other: 6. Fish and soda, no meat
- 7. No meat, fish, or soda (Experimental): no fish, and no soda (vegetarian) for 12 weeks
  Interventions: Other: 7. No meat, fish or soda
- 8. Soda, no meart or fish (Experimental): weight maintaining diet with soda but no meat or fish (vegetarian + soda) for 12 weeks
  Interventions: Other: 8. Soda, no meat or fish
- Meat and fish, no soda (Experimental): weight maintaining diet with meat and fish but no soda for 12 weeks
  Interventions: Other: 3. Meat and fish, no soda

INTERVENTIONS:
Other: 1. Meat, no fish or soda — weight maintaining diet with meat but no fish or soda
  Arms: 1. Meat, no fish or soda
Other: 2. Meat and soda, no fish — weight maintaining diet with meat and soda but no fish
  Arms: 2. Meat and soda, no fish
Other: 3. Meat and fish, no soda — weight maintaining diet with meat and fish but no soda
  Arms: Meat and fish, no soda
Other: 4. Meat and fish and soda — weight maintaining diet with meat, fish and soda
  Arms: 4. Meat and fish and soda
Other: 5. Fish, no meat or soda — weight maintaining diet with fish but no meat or soda
  Arms: 5. Fish, no meat or soda
Other: 6. Fish and soda, no meat — weight maintaining diet with fish and soda but no meat
  Arms: 6. Fish and soda, no meat
Other: 7. No meat, fish or soda — weight maintaining diet with no meat, no fish, and no soda (vegetarian)
  Arms: 7. No meat, fish, or soda
Other: 8. Soda, no meat or fish — weight maintaining diet with soda but no meat or fish (vegetarian + soda)
  Arms: 8. Soda, no meart or fish

SUMMARY:
Background:

- Researchers who study health and nutrition are interested in developing more accurate methods of determining what people eat from day to day and how it affects their general health. In particular, better methods are needed to determine if people are accurately remembering what they ate. One possible method involves the use of biomarkers, or indicators in urine, blood, saliva, fat, and hair, which are related to the intake of a particular food in a consistent way. One set of biomarkers in blood samples and hair may be used to determine the relative amount of meat, fish, and soda (corn/sugar cane) in a person s diet. However, more research is needed to study the effectiveness of using these biomarkers to accurately track dietary intake.

Objectives:

- To validate the use of biomarkers as representative of specific dietary intake patterns (meat/fish/soda).

Eligibility:

- Healthy, nondiabetic men between 18 and 65 years of age.

Design:

* This study involves an initial screening visit and a 12-13 week inpatient dietary study period.
* Participants will be screened with a medical history and physical examination, as well as blood and urine samples and a glucose tolerance test to exclude individuals who have diabetes.
* After 3 days of a standard weight-maintaining diet, participants will have a glucose tolerance test and a body fat scan; provide hair, blood, and fat tissue samples; and complete questionnaires and performance tests.
* Participants will spend one day in a metabolic chamber to measure their energy expenditure and general metabolism.
* Participants will then be randomized into one of eight carefully designed diets for 12 weeks. The diets will differ in the amount of meat, fish, and soda, including one diet where none of the three biomarker-related foods will be permitted. Blood samples will be collected throughout the study diet period.
* At the end of the 12-week study diet period, participants will provide additional hair, blood, and fat tissue samples, and will have a second metabolism assessment in the metabolic chamber....

DETAILED DESCRIPTION:
Studies of health and nutrition use a variety of tools to determine what people eat from day to day. Unfortunately, most of the methods used are not accurate for a variety of reasons and do not provide solid information on which to base health recommendations or public policy. In general, when people are asked to keep track of what they eat or recall what they have eaten in the past, they make mistakes in estimating both amounts and specifics of what was eaten. New tools that can help determine if people are accurately remembering what they ate are desperately needed.

Biomarkers are things that can be measured (in urine, blood, hair, etc.) which are related to the intake of a particular food in a consistent way and may therefore be more accurate than a food record. One set of biomarkers that may be used are naturally occurring (present in all foods) stable isotopes of carbon and nitrogen to determine the relative amount of meat, fish, and soda (corn/sugar cane) in a person s diet. These isotopes can be measured in blood samples and hair.

The aim of this study is to validate the use of stable isotope biomarkers as representative of specific dietary intake patterns (meat/fish/soda). This study will be an inpatient study in which highly specific diets will be fed to volunteers for ~12 weeks and stable isotopes will be measured in blood and hair. The ultimate goal is to develop biomarkers to be used to validate food intake patterns in outpatient clinical and epidemiological studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Body mass index less than or equal to 35 kg/m(2) to minimize the impact of body size on isotope measurements.
* Males 18-65 years old will be recruited for this study. Minors under the age of 18 will be excluded because the time requirements of the study are such that they would interfere with school schedules.

Healthy, as determined by medical history, physical examination, and laboratory tests.

EXCLUSION CRITERIA:

* Current smoking
* Female sex
* Baldness or hair less than 2 cm in length
* Medically- or self-imposed dietary restrictions that would limit a participant s ability/willingness to consume the diet to which they are randomized.
* Type 2 diabetes (according to the World Health Organization diagnostic criteria)
* Endocrine disorders (Cushing s Disease, pituitary disorders, and hypo- and hyperthyroidism)
* Chronic pulmonary disorders, including chronic obstructive pulmonary disease, that would limit ability to follow the protocol (investigator judgment) and obstructive sleep apnea syndrome; only subjects with mild or exercise-induced asthma on no medications or on beta-adrenergic agonists only (such as albuterol) will be allowed to enter the study (provided use of these agents is not required for one week before study entry).
* Cardiovascular diseases (coronary heart disease, heart failure, arrhythmias, and peripheral artery disease)
* Hypertension (blood pressure measurement higher than 140/90 mm Hg on two or more occasions or use of anti-hypertensive medications)
* Diagnosed gastrointestinal diseases, including inflammatory bowel diseases (e.g., Crohn s disease and ulcerative colitis), malabsorption syndromes (e.g., celiac disease), gastric ulcer (active); only subjects with gastro-esophageal reflux will be allowed to enter the study
* Presence of a pacemaker or other implantable devices
* Liver disease (cirrhosis, active hepatitis B or C, and AST or ALT greater than or equal to 1.5 x normal)
* Renal disease (serum creatinine concentrations greater than or equal to 1.5 mg/dl and/or greater than 100mg/dl of protein based on urine dipstick)
* Central nervous system disease (cerebrovascular accidents, dementia, and neurodegenerative disorders)
* Cancer requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis
* Alcohol (more than 3 drinks per day) and/or drug abuse (such as amphetamines, cocaine, heroin, or marijuana)
* Current or past history of: bipolar disorder, schizophrenia or presence of psychotic symptoms, bulimia nervosa or anorexia nervosa, or current major depressive disorder
* Weight change of plus or minus 5% in the last 3 months

Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the investigators. Additionally, potential subjects might be excluded if they demonstrate a style of interpersonal relationships that would inhibit successful completion of the study.

Non-English speaking subjects as a population will be excluded from participation in this protocol. One of the secondary hypotheses of the protocol relates to a battery of psychological questionnaires and performances tests which are administered to the volunteers at the beginning and end of the study. There are currently no validated, translated forms of these questionnaires and tests available; therefore we will restrict enrollment to English speaking subjects only.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-10-24; Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in NIR | Weeks 0, 2, 4, 6, 8, 10, 12
  Change in nitrogen stable isotope rations (N15/N14)
Change in CR | Weeks 0, 2, 4, 6, 8, 10, 12
  Change in carbon stable isotope ratios (13C/12C)

SECONDARY OUTCOMES:
Performance tests | Weeks 0 and 12
  Iowa Card Setting Test, Stroop Color Word Test, Wisconsin Card Sorting Test, Go/No Go Task
OGTT | Weeks 0 and 12
Lipid panel | Weeks 0 and 12
  LDL, HDL, Triglycerides and Total Cholesterol
Respiratory quotient (RQ) | Weeks 0 and 12
  Ratio of the volume of carbon dioxide (CO2) produced to the volume of oxygen (O2) used, or VCO2/VO2

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Votruba, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Kipnis V, Subar AF, Midthune D, Freedman LS, Ballard-Barbash R, Troiano RP, Bingham S, Schoeller DA, Schatzkin A, Carroll RJ. Structure of dietary measurement error: results of the OPEN biomarker study. Am J Epidemiol. 2003 Jul 1;158(1):14-21; discussion 22-6. doi: 10.1093/aje/kwg091. PMID 12835281
- [Background] Subar AF, Kipnis V, Troiano RP, Midthune D, Schoeller DA, Bingham S, Sharbaugh CO, Trabulsi J, Runswick S, Ballard-Barbash R, Sunshine J, Schatzkin A. Using intake biomarkers to evaluate the extent of dietary misreporting in a large sample of adults: the OPEN study. Am J Epidemiol. 2003 Jul 1;158(1):1-13. doi: 10.1093/aje/kwg092. PMID 12835280
- [Background] Tarasuk V, Beaton GH. The nature and individuality of within-subject variation in energy intake. Am J Clin Nutr. 1991 Sep;54(3):464-70. doi: 10.1093/ajcn/54.3.464. PMID 1877501
- [Derived] Johnson JJ, Ghosh S, Shaw PA, Neuhouser ML, Lampe JW, Tinker LF, Prentice RL, Tasevska N, Freedman LS, Boyer BB, Hopkins SE, Nash SH, Votruba SB, Krakoff J, O'Brien DM. The carbon isotope ratio of alanine is a biomarker of added sugar and sugar-sweetened beverage intakes: a pooled analysis of 4 studies. Am J Clin Nutr. 2025 Dec;122(6):1769-1777. doi: 10.1016/j.ajcnut.2025.09.049. Epub 2025 Oct 3. PMID 41047130
- [Derived] Mitchell CM, Oxtoby LE, Shaw PA, Budge SM, Wooller MJ, Cabeza de Baca T, Krakoff J, Votruba S, O'Brien DM. Carbon Isotope Ratios of Plasma and RBC Fatty Acids Identify Meat Consumers in a 12-Week Inpatient Feeding Study of 32 Men. J Nutr. 2023 Jan 14;152(12):2847-2855. doi: 10.1093/jn/nxac213. PMID 36095134
- [Derived] Johnson JJ, Shaw PA, Wooller MJ, Venti CA, Krakoff J, Votruba SB, O'Brien DM. Amino Acid Nitrogen Isotope Ratios Respond to Fish and Meat Intake in a 12-Week Inpatient Feeding Study of Men. J Nutr. 2022 Sep 6;152(9):2031-2038. doi: 10.1093/jn/nxac101. PMID 35511610
- [Derived] Mitchell CM, Piaggi P, O'Brien DM, Krakoff J, Votruba SB. Metabolic Characterization of Meat, Fish, and Soda Intake in Males: Secondary Results from a Randomized Inpatient Pilot Study. Obesity (Silver Spring). 2021 Jun;29(6):995-1002. doi: 10.1002/oby.23167. Epub 2021 May 3. PMID 33938613
- [Derived] Johnson JJ, Shaw PA, Oh EJ, Wooller MJ, Merriman S, Yun HY, Larsen T, Krakoff J, Votruba SB, O'Brien DM. The carbon isotope ratios of nonessential amino acids identify sugar-sweetened beverage (SSB) consumers in a 12-wk inpatient feeding study of 32 men with varying SSB and meat exposures. Am J Clin Nutr. 2021 May 8;113(5):1256-1264. doi: 10.1093/ajcn/nqaa374. PMID 33676366
- [Derived] Votruba SB, Shaw PA, Oh EJ, Venti CA, Bonfiglio S, Krakoff J, O'Brien DM. Associations of plasma, RBCs, and hair carbon and nitrogen isotope ratios with fish, meat, and sugar-sweetened beverage intake in a 12-wk inpatient feeding study. Am J Clin Nutr. 2019 Dec 1;110(6):1306-1315. doi: 10.1093/ajcn/nqz208. PMID 31515553
- [Derived] Stinson EJ, Graham AL, Thearle MS, Gluck ME, Krakoff J, Piaggi P. Cognitive dietary restraint, disinhibition, and hunger are associated with 24-h energy expenditure. Int J Obes (Lond). 2019 Jul;43(7):1456-1465. doi: 10.1038/s41366-018-0305-9. Epub 2019 Jan 16. PMID 30651576